CLINICAL TRIAL: NCT06045949
Title: Prediction of Early Recovery of Liver Function After Living Donor Liver Transplantation in Children: An Ambispective Cohort Study
Brief Title: Prediction of Early Recovery of Liver Function After LDLT in Children: An Ambispective Cohort Study
Status: Completed | Type: Observational
Sponsor: Huiwu Xing (Other)
Responsible Party: Sponsor-Investigator, Huiwu Xing, Dr., Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Other Study IDs: DRHFafterLDLT
Record Dates: First submitted 2023-09-09; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Liver and Biliary Tract Disorders in Duration of Pregnancy; Other End-stage Liver Diseases in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- living donor liver transplantation in children

SUMMARY:
The investigators included children with living donor liver transplantation (LDLT) from January 1, 2018 to July 31, 2022 as a retrospective cohort, and the group from August 1, 2022 to June 30, 2023 as a prospective cohort. The investigators collected the demographic and clinicopathological data of donors and recipients, and determined the risk factors of early postoperative delayed recovery of hepatic function (DRHF) by univariate and multivariate Logical regression analyses.

ELIGIBILITY:
Inclusion Criteria:

1. children with the indication of LDLT [cholestatic liver disease (such as BA), metabolic liver disease (such as Wilson's disease and Ornithine transcarbamylase deficiency), acute liver failure (such as drug induced), neoplastic disease (such as hepatoblastoma), vascular disease (such as cavernous transformation of portal vein and congenital absence of portal vein), re-transplantation and others];
2. the relatives of the children voluntarily donated part of the liver which met the requirements of LDLT.

Exclusion Criteria:

1. recipients with contraindications of LDLT (such as coagulation dysfunction, acute infection, cardiopulmonary failure);
2. failure to complete LDLT due to various reasons (such as death during or within 3 days after operation);
3. recipients or donors with incomplete necessary data.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The investigators included children who underwent LDLT in this center from January 1, 2018 to June 30, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2022-07-31 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
DRHF | 30 days after LDLT in children
  Investigators collected liver function data of children after LDLT. Delayed recovery of hepatic function (DRHF) is characterized by the increase of PT-INR combined with hyperbilirubinemia on or after postoperative day 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No